CLINICAL TRIAL: NCT03512197
Title: A Phase III, Randomized, Double-blind Study of Chemotherapy With Daunorubicin or Idarubicin and Cytarabine for Induction and Intermediate Dose Cytarabine for Consolidation Plus Midostaurin (PKC412) or Chemotherapy Plus Placebo in Newly Diagnosed Patients With FLT-3 Mutation Negative Acute Myeloid Leukemia (AML)
Brief Title: A Global Study of the Efficacy and Safety of Midostaurin + Chemotherapy in Newly Diagnosed Patients With FLT3 Mutation Negative (FLT3-MN) Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPKC412E2301; 2017-003540-21 (EudraCT Number)
Record Dates: First submitted 2018-03-26; First posted 2018-04-30 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Newly diagnosed FLT3-mutation negative; PKC412; midostaurin; cytarabine; daunorubicin; idarubicin; acute myeloid leukemia; AML; FLT3-MN (SR<0.05); combination treatment; induction failure; event free survival; EFS; minimal residual disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — midostaurin; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Midostaurin + chemotherapy (Experimental): Participants received Midostaurin in Induction 50mg twice daily on Day 8 until 48 hrs before start of next cycle. During Induction 2 and consolidation 50mg twice daily on Day 4 until 48 hrs before start of next cycle. During post-consolidation 50mg twice daily for 28 consecutive days of each 28-day treatment cycle up to 12 cycles. For participants who could not tolerate the protocol-specified dosing schedule, dose interruptions and/or reductions were either recommended or mandated allowing participants to continue the study treatment. Chemotherapy consisted of daunorubicin or idarubicin and cytarabine for induction and intermediate dose cytarabine for consolidation.
  Interventions: Drug: Midostaurin; Drug: Chemotherapy
- Placebo + chemotherapy (Placebo Comparator): Participants received matching placebo to midostaurin with same dose, plus chemotherapy. Chemotherapy consisted of daunorubicin or idarubicin and cytarabine for induction and intermediate dose cytarabine for consolidation
  Interventions: Drug: Placebo; Drug: Chemotherapy

INTERVENTIONS:
Drug: Midostaurin — Midostaurin was provided as 25 mg capsules 8PC, was supplied as double-blind in blister packs and taken orally.
  Other Names: PKC412
  Arms: Midostaurin + chemotherapy
Drug: Placebo — Placebo was provided as 25 mg soft gelatin capsules 8PC, was supplied as double-blind in blister packs and taken orally.
  Arms: Placebo + chemotherapy
Drug: Chemotherapy — Along with the study drug/placebo, chemotherapy was given as well: either Daunorubicin or Idarubicin and Cytarabine - all taken by i.v.

SUMMARY:
The purpose of this study was to confirm the preliminary evidence from early clinical trials that midostaurin may provide clinical benefit not only to AML patients with the FLT3-mutations but also in FLT3-MN (SR<0.05) AML (FLT3 mutant to wild type signal ratio below the 0.05 clinical cut-off).

This study evaluated the efficacy and safety of midostaurin in combination with daunorubicin or idarubicin and cytarabine for induction and intermediate-dose cytarabine for consolidation, and midostaurin single agent post-consolidation therapy in newly diagnosed patients with FLT3-MN (SR<0.05) AML.

DETAILED DESCRIPTION:
This was a multi-center, multinational, randomized, double-blind Phase III study using a group sequential design. Subjects were stratified according to age (<60 vs. ≥ 60 years). Subjects within each stratum were randomized in a 1:1 ratio into one of two treatment arms: Midostaurin + chemotherapy 'or' Placebo + chemotherapy.

The study consisted of the following phases:

Screening/randomization phase: Subjects had to sign informed consent form before screening for enrollment. Subjects started chemotherapy at day 1 and were randomized at day 8.

Induction phase: All subjects received at least one cycle (28 days) of induction therapy with continuous infusion cytarabine (D1 - D7) and daunorubicin or idarubicin (D1 - D3) (induction 1). Subjects who did not achieve CR or CRi with adequate blood count recovery after Induction 1 received a second cycle with intermediate-dose cytarabine (D1 - D3) and daunorubicin or idarubicin (D1 - D3) (induction 2). Subjects who did not achieve CR or CRi with adequate blood recovery after induction 2 discontinued study treatment and were followed for survival.

Consolidation phase: Subjects who achieved CR or CRi with adequate blood count recovery after induction with one or two cycles of induction proceeded to consolidation therapy with either 3 or 4 cycles respectively of intermediate-dose cytarabine (D1 - D3), or to Hematopoietic Stem Cells Transplantation (HSCT) with or without preceding consolidation cycles.

Post-consolidation phase: Subjects who maintained CR or CRi with adequate blood count recovery at the end of the consolidation phase received 12 cycles (28 days/cycle) of continuous therapy with midostaurin or placebo twice daily at 50 mg. Subjects who underwent HSCT after achieving CR or CRi with adequate blood count recovery received midostaurin or placebo twice daily 50 mg post-transplant therapy, continuously, for up to 12 cycles (28 days/cycle). Post HSCT post-consolidation therapy began >30 days but not later than 100 days following HSCT.

Follow-up phase: All enrolled subjects were followed through the treatment period and until relapse/treatment failure, thereafter for start of new line of therapy and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AML (≥20% blasts in the bone marrow based on WHO 2016 classification). Patients with APL with PML-RARA are not eligible.
2. Suitability for intensive induction chemotherapy in the judgment of the investigator
3. Documented absence of an ITD and TKD activating mutation at codons D835 and I836 in the FLT3 gene, as determined by analysis in a Novartis designated laboratory using a validated clinical trial assay with clinical cutoff of 0.05 mutant to wild type signal ratio
4. Age ≥18 years
5. Laboratory values that indicate adequate organ function assessed locally at the screening visit

Exclusion Criteria:

1. Central nervous system (CNS) leukemia
2. Therapy-related secondary AML
3. Isolated extramedullary leukemia
4. Prior therapy for leukemia or myelodysplasia
5. AML after antecedent myelodysplasia (MDS) with prior cytotoxic treatment (e.g., azacytidine or decitabine)
6. Prior treatment with a FLT3 inhibitor (e.g., midostaurin, quizartinib, sorafenib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (124):
- United States (3):
  - University of Chicago Medical Center ., Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Oregon Health and Science Univ, Portland, Oregon
- Novartis Investigative Site, CABA, Buenos Aires, Argentina
- Australia (4):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Prahran, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
- Austria (2):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (3):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Roeselare
- Brazil (3):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São Paulo
- Novartis Investigative Site, Sofia, Bulgaria
- Czechia (2):
  - Novartis Investigative Site, Brno-Bohunice
  - Novartis Investigative Site, Plzen-Bory
- France (9):
  - Novartis Investigative Site, Bayonne, Bayonne Cedex
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Toulouse
- Germany (33):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Schwerin, Brandenburg
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eschweiler
  - Novartis Investigative Site, Essen Werden
  - Novartis Investigative Site, Flensburg
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Paderborn
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Würzburg
  - Novartis Investigative Site, Zwickau
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv
- Italy (16):
  - Novartis Investigative Site, Alessandria, AL
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Piacenza, PC
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Taranto, TA
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Vicenza, VI
- Japan (20):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Fukuyama, Hiroshima
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Aomori
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Yamagata
- Norway (2):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo
- Novartis Investigative Site, Gdansk, Poland
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Spain (10):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barakaldo, Basque Country
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich
- Taiwan (4):
  - Novartis Investigative Site, Putzu City, Chiayi Hsien
  - Novartis Investigative Site, Kuei Shan Chiang, Taoyuan Taiwan ROC
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Aydin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five hundred and three participants were randomized. However, 2 patients were randomized by error and got discontinued right after randomization. Therefore, the data analysis was considered for 501 participants only (250 participants in midostaurin arm and 251 participants in placebo arm).
Pre-assignment Details: Participants had to sign informed consent form before screening for enrollment. Participants started chemotherapy at day 1 and were randomized at day 8.
Period: Overall Study
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Started (Randomized) | 250 | 251
Treated With Midostaurin/Placebo | 245 | 249
Entered Induction Phase | 250 | 251
Entered Consolidation Phase | 120 | 129
Entered Post-Consolidation Phase | 45 | 27
Completed (Completed entire study treatment as per protocol - defined as completion of induction, consolidation and post-consolidation treatment phases) | 2 | 1
Not Completed | 248 | 250
Not completed — Guardian decision | 1 | 1
Not completed — Lack of Efficacy | 19 | 11
Not completed — New Therapy for Study Indication | 16 | 16
Not completed — Physician Decision | 60 | 60
Not completed — Protocol Violation | 0 | 2
Not completed — Terminated by Sponsored | 46 | 50
Not completed — Subject Decision | 15 | 12
Not completed — Withdrawal of informed consent | 20 | 14
Not completed — Adverse Event | 30 | 34
Not completed — Death | 14 | 9
Not completed — Failure to meet Continuation Criteria | 24 | 28
Not completed — Missing | 3 | 13

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) comprised all participants to whom study drug was assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy | Total
Number analyzed (Participants) | 250 | 251 | 501
Age, Continuous [Median (Full Range); unit: Years] | 58.0 [19.0 to 78.0] | 58.0 [18.0 to 79.0] | 58.0 [18.0 to 79.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 106 | 228
  Male | 128 | 145 | 273
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 213 | 208 | 421
  Black or African American | 1 | 2 | 3
  Asian | 22 | 22 | 44
  Multiple | 1 | 1 | 2
  Missing | 13 | 18 | 31
ECOG performance status [Count of Participants; unit: Participants] — ECOG performance status determines the ability of a patient to tolerate therapies in serious illness, specifically for chemotherapy.
  Participants
    0 (Asymptomatic) | 119 | 119 | 238
    1 (Symptomatic, fully ambulatory) | 107 | 115 | 222
    2 (Symptomatic, in bed <50% of the day) | 18 | 13 | 31
    3 (Symptomatic, in bed >50% of the day) | 2 | 0 | 2
    Missing | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival (EFS)
Description: EFS was defined as the time from randomization to failure to obtain a complete remission (CR) or Complete remission with incomplete hematologic recovery (CRi) with adequate blood count recovery in induction, relapse after CR or CRi with adequate blood count recovery or death due to any cause, whichever occurred first as assessed by the investigator.
Time Frame: From date of Randomization up to approx. 30 months
Population: Full analysis set comprised all participants to whom study drug was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 250 | 251
Months | 5.98 [2.33 to 8.97] | 5.88 [3.65 to 7.52]
Statistical Analysis 1: Comparison: Midostaurin + Chemotherapy vs Placebo + Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 1.0239, 95% CI 2-sided [0.8 to 1.31]

2. Secondary Outcome: Overall Survival (OS) (Key Secondary)
Description: OS was defined as the time from randomization to date of death due to any cause. Patients entered the survival follow-up phase once they completed the safety follow up period (30 days after the last dose of midostaurin/placebo) in case of induction failure or if they had relapsed during post-treatment follow-up. Patients were then contacted by telephone every 3 months +/- 2 weeks or had a visit to follow up on their survival status, per Kaplan-Meier estimates.
Time Frame: Between randomization to date of death up to approx. 30 months
Population: Full analysis set comprised all participants to whom study drug was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 250 | 251
Months | NA [15.54 to NA] — N/A: Very low number of OS events did not allow to estimate median of OS nor the boundaries of CI. Study was stopped at first interim analysis and thus the survival follow-up was stopped also. | 19.22 [13.8 to NA] — N/A: Very low number of OS events did not allow to estimate the boundaries of CI. Study was stopped at first interim analysis and thus the survival follow-up was stopped also.
Statistical Analysis 1: Comparison: Midostaurin + Chemotherapy vs Placebo + Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.8728, 95% CI 2-sided [0.59 to 1.29]

3. Secondary Outcome: Percentage of Participants With Complete Remission (CR) and Complete Remission With Incomplete Hematological Recovery (CRi) But With Adequate Blood Count Recovery Rate.
Description: Assessment was based on the International Working Group (IWG) criteria for AML as per investigator assessment.
  CR: Bone marrow: < 5% blasts no blasts with Auer rods; Peripheral blood: neutrophils ≥ 1.0 x 109/L platelets ≥ 100 x 109/L, no blasts; No evidence of extramedullary disease (such as central nervous system (CNS) or soft tissue involvement); Transfusion independent.
  CRi with adequate blood count recovery is defined as the following:
  Bone marrow < 5% blasts no blasts with Auer rods Peripheral blood Neutrophils >= 1.0 x 109/L and 50 x 109/L <=platelets < 100 x 109/L no blasts No evidence of extramedullary disease (such as CNS or soft tissue involvement).
Time Frame: At maximum 93 days from induction therapy start
Population: Full analysis set comprised all participants to whom study drug was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 250 | 251
Percentage of participants | 59.2 [52.8 to 65.4] | 61.0 [54.6 to 67.0]

4. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD) Negative Status
Description: MRD- rate was defined as the rate of participants reaching MRD at any timepoint. Participants with leukemic blasts below 0.1% were considered as MRD-negative based on leukemia-associated immunophenotype (LAIP).
  MRD was derived from bone marrow and blood data using cellular and molecular technologies and MRD status was measured using the flow cytometry assessments for LAIP irrespective of the investigator's overall clinical response assessment.
Time Frame: from start of treatment up to end of post-consolidation (approximately 17 months)
Population: Full analysis set comprised all participants to whom study drug was assigned by randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 250 | 251
Percentage of participants | 40.8 | 41.0

5. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD) Negative Status During Post-consolidation Phase
Description: MRD- rate was defined as the rate of participants reaching MRD at any timepoint during Post-consolidation phase. Participants with leukemic blasts below 0.1% were considered as MRD-negative based on leukemia-associated immunophenotype (LAIP).
  MRD was derived from bone marrow and blood data using cellular and molecular technologies and MRD status was measured using the flow cytometry assessments for LAIP irrespective of the investigator's overall clinical response assessment.
Time Frame: from start of post-consolidation to end of post-consolidation phase (up to 12 months)
Population: Full analysis in post-consolidation phase comprised of participants who entered post-consolidation phase
Measure: Number; unit: Percentage of participants
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 45 | 27
Percentage of participants | 33.3 | 33.3

6. Secondary Outcome: Time to Measurable Residual Disease (MRD) Negativity by Flow Cytometry
Description: Time to MRD- is defined as time from randomization to first occurrence of MRD-. Participants with leukemic blasts below 0.1% were considered as MRD-negative based on leukemia-associated immunophenotype (LAIP).
  MRD was derived from bone marrow and blood data using cellular and molecular technologies and MRD status was measured using the flow cytometry assessments for LAIP irrespective of the investigator's overall clinical response assessment.
Time Frame: From date of Randomization up to approx. 17 months
Population: Analysis set comprised all participants to whom study drug was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 250 | 251
Days | 2.27 [1.61 to 5.68] | 2.07 [1.68 to 6.80]

7. Secondary Outcome: Disease-free Survival (DFS)
Description: DFS as measured from the date of first CR or CRi with adequate blood count recovery to relapse or death due to any cause, whichever occurred first. Participants who did not relapse nor die were censored at the last adequate response assessment. Assessment was based on the IWG criteria for AML as per investigator assessment
Time Frame: From date of CR or CRi with adequate blood count recovery up to approx. 30 months
Population: Full analysis set comprised all participants to whom study drug was assigned by randomization. DFW was derived only for participants who reached CR or CRi with adequate blood count recovery in induction (during first 93 days).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 148 | 153
Months | 10.5 [7.59 to NA] — N/A: Upper limit of CI could not be reached because of low number of events due to premature study discontinuation | 9.1 [6.87 to 12.02]
Statistical Analysis 1: Comparison: Midostaurin + Chemotherapy vs Placebo + Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.60 to 1.63]

8. Secondary Outcome: Cumulative Incidence of Relapse (CIR)
Description: Cumulative Incidence of Relapse (CIR) was defined for participants with CR or CRi with adequate blood count recovery and was the time from achieving the CR or CRi with adequate blood count recovery until the onset of relapse from CR or CRi with adequate blood recovery. Participants without relapse were censored at the last adequate response assessment. Participants who died without relapse were counted as a competing cause of failure.
Time Frame: From date of CR or CRi with adequate blood count recovery up to approx. 30 months
Population: Full analysis set comprised all participants to whom study drug was assigned by randomization. CIR was only for participants who achieved CR or CRi with adequate blood count recovery.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 148 | 153
Months | 5.1 [2.83 to 7.56] | 6.6 [4.99 to 8.77]
Statistical Analysis 1: Comparison: Midostaurin + Chemotherapy vs Placebo + Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 1.5866, 95% CI 2-sided [0.88 to 2.87]

9. Secondary Outcome: Cumulative Incidence of Death (CID)
Description: Cumulative Incidence of Death (CID) was defined for all participants achieving CR or CRi with adequate blood count recovery measured from the date of achievement of CR or CRi until the date of death due to any reason. Participants not known to have died were censored on the last contact date. Participants who experienced relapse were counted as a competing cause of failure.
Time Frame: From date of CR or CRi with adequate blood count recovery up to approx. 30 months
Population: Full analysis set comprised all participants to whom study drug was assigned by randomization. CID was only for participants who achieved CR or CRi with adequate blood count recovery.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 148 | 153
Months | NA [18.00 to NA] — N/A: Very low number of events did not allow to estimate median of CID nor the boundaries of CI. | NA [14.42 to NA] — N/A: Very low number of events did not allow to estimate median of CID nor the boundaries of CI
Statistical Analysis 1: Comparison: Midostaurin + Chemotherapy vs Placebo + Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.7937, 95% CI 2-sided [0.41 to 1.54]

10. Secondary Outcome: Time to CR or CRi With Adequate Blood Count Recovery
Description: Time to CR or CRi with adequate blood count recovery was defined as the time from randomization to CR or CRi with adequate blood count recovery whichever occurred first
Time Frame: At maximum 93 days from induction therapy start
Population: Full analysis set comprised all participants to whom study drug was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 250 | 251
Days | 1.12 [1.02 to 1.41] | 1.15 [1.05 to 1.54]

11. Secondary Outcome: Time to Partial and Full Neutrophil Recovery
Description: The time to neutrophil recovery was assessed for the following criteria: Partial neutrophil recovery: Number of days from start of treatment to the first day neutrophils ≥0.5 x 10^9/L.
  Full neutrophil recovery: Number of days from start of treatment to the first day neutrophils ≥1.0 x 10^9/L
Time Frame: At maximum 93 days from induction therapy start
Population: Full analysis set comprised all participants to whom study drug was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 250 | 251
Months
  Partial neutrophil recovery | 1.1 [0.82 to 1.15] | 0.9 [0.79 to 1.12]
  Full neutrophil recovery | 1.2 [1.05 to 1.48] | 1.1 [0.95 to 1.35]
Statistical Analysis 1: Comparison: Midostaurin + Chemotherapy vs Placebo + Chemotherapy; partial neutrophil recovery; Test type: Superiority; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.75 to 1.16]
Statistical Analysis 2: Comparison: Midostaurin + Chemotherapy vs Placebo + Chemotherapy; full neutrophil recovery; Test type: Superiority; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.72 to 1.14]

12. Secondary Outcome: Time to Partial and Full Platelet Recovery
Description: Time to platelet recovery was assessed for the following criteria: Partial platelet recovery: Number of days from start of treatment to the first day platelets ≥50 x 10^9/L.
  Full platelet recovery: Number of days from start of treatment to the first day platelets ≥100 x 10^9/L.
Time Frame: At maximum 93 days from induction therapy start
Population: Full analysis set comprised all participants to whom study drug was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 250 | 251
Months
  Partial platelet recovery | NA [1.45 to NA] — N/A: Very low number of events did not allow to estimate median nor the boundaries of CI. | NA [3.5 to NA] — N/A: Very low number of events did not allow to estimate median nor the boundaries of CI.
  Full platelet recovery | 0.953 [0.89 to 1.12] | 0.887 [0.85 to 0.92]
Statistical Analysis 1: Comparison: Midostaurin + Chemotherapy vs Placebo + Chemotherapy; partial platelet recovery; Test type: Superiority; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.87 to 1.52]
Statistical Analysis 2: Comparison: Midostaurin + Chemotherapy vs Placebo + Chemotherapy; full platelet recovery; Test type: Superiority; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.67 to 1.00]

13. Secondary Outcome: Plasma Concentrations for Midostaurin and Its Metabolites: CGP52421 and CGP62221 for Non-poor Metabolizers
Description: Serial pharmacokinetics (PK) samples were collected in Non-poor metabolizer participants to assess the plasma concentrations of midostaurin, CGP52421 and CGP62221.
Time Frame: from Induction (IND) phase 0hr (predose) to Post-consolidation phase (POSTCONS) 12hr
Population: Pharmacokinetic analysis set-all (PAS-all) included all participants in the safety set who provided at least one evaluable PK concentration for Non-poor metabolizers. PK samples were not collected in all timepoints of all patients and reported for Non-poor metabolizers only.
Measure: Mean (Standard Deviation); unit: hour (hr)
Groups:
- CGP52421; CGP62221: Active Midostaurin metabolite
Arm/Group | Midostaurin + Chemotherapy | CGP52421 | CGP62221
Number analyzed (Participants) | 145 | 145 | 145
hour (hr)
  IND C1D8 0hr (Predose) (n = 34, 34, 34): number analyzed (Participants) | 34 | 34 | 34
  IND C1D8 0hr (Predose) (n = 34, 34, 34) | 0 (0) | 0 (0) | 0 (0)
  IND C1D8 1hr (n= 6, 6, 6): number analyzed (Participants) | 6 | 6 | 6
  IND C1D8 1hr (n= 6, 6, 6) | 1110 (791) | 30.0 (35.4) | 37.6 (45.3)
  IND C1D8 3hr (n = 108, 104, 108): number analyzed (Participants) | 108 | 104 | 108
  IND C1D8 3hr (n = 108, 104, 108) | 2000 (897) | 80.6 (48.8) | 198 (178)
  IND C1D8 6hr ( n= 7, 7, 7): number analyzed (Participants) | 7 | 7 | 7
  IND C1D8 6hr ( n= 7, 7, 7) | 1370 (448) | 92.1 (47.1) | 285 (222)
  IND C1D8 12hr (n= 7, 7, 7): number analyzed (Participants) | 7 | 7 | 7
  IND C1D8 12hr (n= 7, 7, 7) | 1090 (365) | 79.3 (31.4) | 280 (196)
  IND C1D11 0hr (Predose) (n = 33, 33, 33): number analyzed (Participants) | 33 | 33 | 33
  IND C1D11 0hr (Predose) (n = 33, 33, 33) | 5340 (3190) | 417 (162) | 1470 (812)
  IND C1D11 3hr (n = 92, 92, 92): number analyzed (Participants) | 92 | 92 | 92
  IND C1D11 3hr (n = 92, 92, 92) | 6840 (3480) | 451 (157) | 1520 (777)
  IND C1D11 12hr (n = 57, 57, 57): number analyzed (Participants) | 57 | 57 | 57
  IND C1D11 12hr (n = 57, 57, 57) | 4800 (2860) | 430 (167) | 1590 (732)
  IND C1D15 0hr (Predose) (n = 25, 25, 25): number analyzed (Participants) | 25 | 25 | 25
  IND C1D15 0hr (Predose) (n = 25, 25, 25) | 8330 (5300) | 776 (261) | 3030 (1460)
  IND C1D15 12hr (n = 63, 63, 63): number analyzed (Participants) | 63 | 63 | 63
  IND C1D15 12hr (n = 63, 63, 63) | 7010 (4260) | 828 (229) | 3170 (1310)
  IND C1D18 0hr (Predose) (n = 19, 19, 19): number analyzed (Participants) | 19 | 19 | 19
  IND C1D18 0hr (Predose) (n = 19, 19, 19) | 6520 (5230) | 1090 (304) | 4070 (1400)
  IND C1D18 12hr (n = 50, 50, 50): number analyzed (Participants) | 50 | 50 | 50
  IND C1D18 12hr (n = 50, 50, 50) | 5960 (4040) | 1050 (332) | 3990 (1580)
  IND C1D21 0hr (Predose) (n = 26, 26, 26): number analyzed (Participants) | 26 | 26 | 26
  IND C1D21 0hr (Predose) (n = 26, 26, 26) | 6190 (4880) | 1310 (467) | 4540 (1950)
  IND C1D21 3hr (n = 89, 89, 89): number analyzed (Participants) | 89 | 89 | 89
  IND C1D21 3hr (n = 89, 89, 89) | 6740 (4390) | 1240 (380) | 4100 (1680)
  IND C1D21 12hr (n = 61, 61, 61): number analyzed (Participants) | 61 | 61 | 61
  IND C1D21 12hr (n = 61, 61, 61) | 5990 (4460) | 1220 (336) | 4320 (1660)
  CONS C1D4 0hr (predose) (n = 16, 15, 16): number analyzed (Participants) | 16 | 15 | 16
  CONS C1D4 0hr (predose) (n = 16, 15, 16) | 72.0 (128) | 922 (246) | 269 (390)
  CONS C1D4 3hr (n = 49, 44, 49): number analyzed (Participants) | 49 | 44 | 49
  CONS C1D4 3hr (n = 49, 44, 49) | 1110 (660) | 1090 (409) | 615 (601)
  CONS C1D4 12hr (n = 2, 2, 2): number analyzed (Participants) | 2 | 2 | 2
  CONS C1D4 12hr (n = 2, 2, 2) | 187 (264) | 1060 (49.5) | 376 (531)
  CONS C1D17 0hr (predose) (n = 14, 14, 14): number analyzed (Participants) | 14 | 14 | 14
  CONS C1D17 0hr (predose) (n = 14, 14, 14) | 1630 (780) | 1860 (387) | 1890 (608)
  CONS C1D17 3hr (n = 48, 47, 48): number analyzed (Participants) | 48 | 47 | 48
  CONS C1D17 3hr (n = 48, 47, 48) | 2580 (1430) | 1620 (505) | 2030 (677)
  CONS C1D17 12hr (n = 29, 29, 29): number analyzed (Participants) | 29 | 29 | 29
  CONS C1D17 12hr (n = 29, 29, 29) | 1950 (1630) | 1710 (500) | 1990 (746)
  CONS C3D4 0hr (predose) ( n = 9, 9, 9): number analyzed (Participants) | 9 | 9 | 9
  CONS C3D4 0hr (predose) ( n = 9, 9, 9) | 94.3 (126) | 968 (469) | 274 (289)
  CONS C3D4 3hr (n = 25, 24, 25): number analyzed (Participants) | 25 | 24 | 25
  CONS C3D4 3hr (n = 25, 24, 25) | 1030 (522) | 983 (465) | 437 (250)
  CONS C3D4 12hr (n = 2, 2, 2): number analyzed (Participants) | 2 | 2 | 2
  CONS C3D4 12hr (n = 2, 2, 2) | 10.6 (14.9) | 996 (105) | 44.1 (41.6)
  CONS C3D17 0hr (predose) (n = 9, 9, 9): number analyzed (Participants) | 9 | 9 | 9
  CONS C3D17 0hr (predose) (n = 9, 9, 9) | 1810 (1470) | 1460 (522) | 1750 (995)
  CONS C3D17 3hr ( n = 24, 24, 24): number analyzed (Participants) | 24 | 24 | 24
  CONS C3D17 3hr ( n = 24, 24, 24) | 2620 (1230) | 1720 (640) | 2140 (1120)
  CONS C3D17 12hr (n = 17, 17, 17): number analyzed (Participants) | 17 | 17 | 17
  CONS C3D17 12hr (n = 17, 17, 17) | 2430 (2450) | 1570 (644) | 1960 (1030)
  POSTCONS C1PRE 0hr (predose) (n = 2, 2, 2): number analyzed (Participants) | 2 | 2 | 2
  POSTCONS C1PRE 0hr (predose) (n = 2, 2, 2) | 472 (407) | 1470 (148) | 786 (487)
  POSTCONS C1PRE 12hr (n = 1, 1, 1): number analyzed (Participants) | 1 | 1 | 1
  POSTCONS C1PRE 12hr (n = 1, 1, 1) | 309 (0) | 1010 (0) | 887 (0)
  POSTCONS C4D1 0hr (predose) (n= 4, 4, 4): number analyzed (Participants) | 4 | 4 | 4
  POSTCONS C4D1 0hr (predose) (n= 4, 4, 4) | 496 (288) | 1070 (396) | 951 (650)
  POSTCONS C4D1 3hr (n = 4, 3, 4): number analyzed (Participants) | 4 | 3 | 4
  POSTCONS C4D1 3hr (n = 4, 3, 4) | 748 (136) | 1180 (458) | 857 (119)
  POSTCONS C4D1 12hr (n = 2, 2, 2): number analyzed (Participants) | 2 | 2 | 2
  POSTCONS C4D1 12hr (n = 2, 2, 2) | 419 (4.95) | 803 (30.4) | 784 (142)
  POSTCONS C7D1 0hr (predose) (n = 1, 1, 1): number analyzed (Participants) | 1 | 1 | 1
  POSTCONS C7D1 0hr (predose) (n = 1, 1, 1) | 311 (0) | 1120 (0) | 896 (0)
  POSTCONS C7D1 12hr (n = 3, 3, 3): number analyzed (Participants) | 3 | 3 | 3
  POSTCONS C7D1 12hr (n = 3, 3, 3) | 639 (174) | 960 (180) | 962 (344)
  POSTCONS C10D1 0hr (predose) (n = 1, 1, 1): number analyzed (Participants) | 1 | 1 | 1
  POSTCONS C10D1 0hr (predose) (n = 1, 1, 1) | 408 (0) | 1020 (0) | 1050 (0)

14. Secondary Outcome: AUC0-t: Pharmacokinetic (PK) Parameter for Midostaurin and Its Metabolites: CGP52421 and CGP62221 at Cycle 1, Day 8
Description: The AUC from time zero to a measurable concentration sampling time (t) (mass x time x volume-1). Note: as the last sampling time was at 12 h, AUC0-12h was determined after the first dose, reported at Cycle 1, Day 8
Time Frame: 0 - 12 hrs
Population: Pharmacokinetic analysis set-all (PAS-all) included all participants in the safety set who provided at least one evaluable PK concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Midostaurin + Chemotherapy | CGP52421 | CGP62221
Number analyzed (Participants) | 20 | 27 | 27
hr*ng/mL | 14800 (37.5) | 712 (78.4) | 1830 (135)

15. Secondary Outcome: AUClast: Pharmacokinetic (PK) Parameter for Midostaurin and Its Metabolites: CGP52421 and CGP62221 at Cycle 1, Day 8
Description: The AUC from time zero to the last measurable concentration sampling time after the first dose reported at Cycle 1, Day 8
Time Frame: 0 - 12 hrs
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Midostaurin + Chemotherapy | CGP52421 | CGP62221
Number analyzed (Participants) | 27 | 27 | 27
hr*ng/mL | 12200 (59.6) | 493 (139) | 1130 (249)

16. Secondary Outcome: Cmax: Pharmacokinetic (PK) Parameter for Midostaurin and Its Metabolites: CGP52421 and CGP62221 at Cycle 1, Day 8
Description: The maximum (peak) observed plasma drug concentration after the first dose administration reported at Cycle 1, Day 8
Time Frame: 0 - 12 hrs
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- GCP62221: Active Midostaurin metabolite
Arm/Group | Midostaurin + Chemotherapy | CGP52421 | GCP62221
Number analyzed (Participants) | 27 | 27 | 27
ng/mL | 1910 (37.8) | 74.7 (72.3) | 183 (128)

17. Secondary Outcome: Tmax: Pharmacokinetic (PK) Parameter for Midostaurin and Its Metabolites: CGP52421 and CGP62221 at Cycle 1, Day 8
Description: The time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after single dose administration reported at Cycle 1, Day 8
Time Frame: 0 - 12 hrs
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (hr)
Groups:
- GCP52421; CGP62221: Active Midostaurin metabolite
Arm/Group | Midostaurin + Chemotherapy | GCP52421 | CGP62221
Number analyzed (Participants) | 27 | 27 | 27
hour (hr) | 3.28 (101) | 5.38 (89.9) | 7.17 (57.8)

18. Secondary Outcome: Total Score for Each Time Point for the Functional Assessment of Cancer Therapy-Leukemia (FACT-Leu)
Description: The total FACT-Leu score consists of 44 items with total scores ranging from 0 to 176. Higher scores indicate better health-related quality of life ( HRQoL). Negative changes from baseline indicate a worsening of HRQoL while positive changes indicate an improvement in HRQoL.
Time Frame: From date of Randomization up to approx. 18 months
Population: Full analysis set comprised all participants to whom study drug was assigned by randomization.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 250 | 251
Scores on a scale
  Baseline (n = 225, 223): number analyzed (Participants) | 225 | 223
  Baseline (n = 225, 223) | 122.8 (22.64) | 123.1 (21.21)
  Induction Phase (n = 137, 147): number analyzed (Participants) | 137 | 147
  Induction Phase (n = 137, 147) | 123.9 (21.50) | 122.1 (19.51)
  Induction I (n = 105, 90): number analyzed (Participants) | 105 | 90
  Induction I (n = 105, 90) | 124.8 (20.34) | 123.5 (20.28)
  Induction ll (n = 32, 57): number analyzed (Participants) | 32 | 57
  Induction ll (n = 32, 57) | 121.0 (25.09) | 119.8 (18.15)
  Consolidation (prior) (n = 210, 196): number analyzed (Participants) | 210 | 196
  Consolidation (prior) (n = 210, 196) | 135.9 (17.67) | 136.9 (21.03)
  Post- consolidation (n = 169, 114): number analyzed (Participants) | 169 | 114
  Post- consolidation (n = 169, 114) | 143.7 (21.45) | 140.1 (21.60)
  Follow-up (n = 74, 111): number analyzed (Participants) | 74 | 111
  Follow-up (n = 74, 111) | 136.4 (22.87) | 139.2 (25.00)

19. Secondary Outcome: Scores for Each Time Point for the EQ5D-5L (a Visual Analogue Scale (VAS))
Description: The EQ5D-5L questionnaire assesses 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response options (no problems, slight problems, moderate problems, severe problems and extreme problems) that reflect increasing levels of difficulty. The patient is asked to indicate his/her current health state by selecting the most appropriate level in each of the 5 dimensions. The questionnaire also included a Visual Analogue Scale (VAS), where the patient is asked to rate current health status on a scale of 0 to 100, with 0 being the worst imaginable health state.
Time Frame: From date of Randomization up to approx. 18 months
Population: Full analysis set comprised all participants to whom study drug was assigned by randomization.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 250 | 251
Scores on a scale
  Baseline ( n= 225, 220): number analyzed (Participants) | 225 | 220
  Baseline ( n= 225, 220) | 62.7 (22.98) | 64.3 (22.15)
  Induction Phase (n = 135, 146): number analyzed (Participants) | 135 | 146
  Induction Phase (n = 135, 146) | 67.9 (20.95) | 64.4 (21.29)
  Induction l (n = 104, 89): number analyzed (Participants) | 104 | 89
  Induction l (n = 104, 89) | 68.1 (21.02) | 64.0 (21.92)
  Induction ll (n = 31, 57): number analyzed (Participants) | 31 | 57
  Induction ll (n = 31, 57) | 66.9 (21.03) | 65.2 (20.44)
  Consolidation (prior) (n = 207, 197): number analyzed (Participants) | 207 | 197
  Consolidation (prior) (n = 207, 197) | 79.1 (15.42) | 76.2 (16.37)
  Post-consolidation (n = 167, 113): number analyzed (Participants) | 167 | 113
  Post-consolidation (n = 167, 113) | 83.9 (15.00) | 77.3 (14.92)
  Follow-up ( n- 74, 112): number analyzed (Participants) | 74 | 112
  Follow-up ( n- 74, 112) | 74.3 (20.08) | 73.4 (1972)

20. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from start of treatment (FPFT) up to 30 days after study drug discontinuation, for a maximum duration of approx. 18 months.
  Randomized but not treated deaths were collected after randomization but before treatment with study drug.
  Post-treatment survival follow-up deaths were collected after the on-treatment period up to approx. 18 months. Participants who did not die during the on-treatment period and had not stopped study participation at the time of data cut-off (when study was terminated) were censored.
Time Frame: Start of study treatment up to 30 days post-treatment for approx. 1 year, prior to study treatment up to LPLV, approx. 18 months
Population: Clinical Database Population: all enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Midostaurin + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 250 | 251
Participants
  Total Deaths | 48 | 54
  Randomized but not treated deaths | 2 | 1
  Deaths on-treatment (n = 245, 249): number analyzed (Participants) | 245 | 249
  Deaths on-treatment (n = 245, 249) | 25 | 21
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 220 | 228
  Post-treatment survival follow-up deaths | 21 | 32

ADVERSE EVENTS:
Time Frame: AEs were reported from 1st dose of study treatment until end of treatment plus 30 days, up to a maximum (max.) duration of 573 days (543 days max. exposure plus 30 days post-treatment) for midostaurin and up to a max. duration of 416 days (386 days max. exp. plus 30 days post-treatment) for placebo. Deaths - collected in the post-treatment survival follow-up period from 31 days after last dose of study medication until the end of the study, up to approx. 18 months. These are not considered AEs.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Deaths in the post-treatment survival follow-up are not considered Adverse Events. The total number at risk in the post-treatment survival includes patients that entered the post-treatment survival follow-up period.
Groups:
- Midostaurin + Chemotherapy (On-treatment); Placebo + Chemotherapy (On-treatment): AEs during on-treatment period (up to 30 days post-treatment)
- Midostaurin + Chemotherapy (Post-treatment Survival Follow-up); Placebo + Chemotherapy (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up phase (starting from day 31 post- treatment). No AEs were collected during this period
Arm/Group | Midostaurin + Chemotherapy (On-treatment) | Placebo + Chemotherapy (On-treatment) | Midostaurin + Chemotherapy (Post-treatment Survival Follow-up) | Placebo + Chemotherapy (Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 25/245 | 21/249 | 21/220 | 32/228
Serious Adverse Events (participants affected / at risk) | 95/245 | 114/249 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 242/245 | 245/249 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Midostaurin + Chemotherapy (On-treatment) (N=245) | Placebo + Chemotherapy (On-treatment) (N=249) | Midostaurin + Chemotherapy (Post-treatment Survival Follow-up) (N=0) | Placebo + Chemotherapy (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 1 | NA | NA
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 1 | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 23 | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | NA | NA
Pancytopenia (Blood and lymphatic system disorders) | 3 | 2 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | NA | NA
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | NA | NA
Atrial fibrillation (Cardiac disorders) | 1 | 3 | NA | NA
Bradycardia (Cardiac disorders) | 0 | 1 | NA | NA
Cardiac arrest (Cardiac disorders) | 1 | 1 | NA | NA
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | NA | NA
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | NA | NA
Myocardial infarction (Cardiac disorders) | 0 | 1 | NA | NA
Myocarditis (Cardiac disorders) | 1 | 0 | NA | NA
Right ventricular dysfunction (Cardiac disorders) | 1 | 0 | NA | NA
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | NA | NA
Aplasia (Congenital, familial and genetic disorders) | 1 | 1 | NA | NA
Thyrotoxic crisis (Endocrine disorders) | 1 | 0 | NA | NA
Anal fistula (Gastrointestinal disorders) | 0 | 1 | NA | NA
Colitis (Gastrointestinal disorders) | 0 | 1 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | NA | NA
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | NA | NA
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | NA | NA
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | NA | NA
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | NA | NA
Jejunal stenosis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 2 | NA | NA
Neutropenic colitis (Gastrointestinal disorders) | 1 | 3 | NA | NA
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1 | NA | NA
Proctalgia (Gastrointestinal disorders) | 1 | 0 | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | NA | NA
Tongue haematoma (Gastrointestinal disorders) | 1 | 0 | NA | NA
Ulcerative duodenitis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Vomiting (Gastrointestinal disorders) | 1 | 2 | NA | NA
Disease progression (General disorders) | 2 | 0 | NA | NA
General physical health deterioration (General disorders) | 0 | 1 | NA | NA
Mucosal inflammation (General disorders) | 1 | 1 | NA | NA
Multiple organ dysfunction syndrome (General disorders) | 2 | 4 | NA | NA
Pyrexia (General disorders) | 4 | 4 | NA | NA
Biliary fistula (Hepatobiliary disorders) | 1 | 0 | NA | NA
Cholecystitis (Hepatobiliary disorders) | 2 | 3 | NA | NA
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1 | NA | NA
Liver disorder (Hepatobiliary disorders) | 0 | 1 | NA | NA
Acute graft versus host disease (Immune system disorders) | 1 | 0 | NA | NA
Anaphylactic reaction (Immune system disorders) | 0 | 1 | NA | NA
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 1 | NA | NA
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0 | NA | NA
Abdominal infection (Infections and infestations) | 1 | 0 | NA | NA
Abscess neck (Infections and infestations) | 1 | 0 | NA | NA
Acinetobacter infection (Infections and infestations) | 0 | 1 | NA | NA
Anal abscess (Infections and infestations) | 1 | 1 | NA | NA
Appendicitis (Infections and infestations) | 0 | 2 | NA | NA
Aspergillus infection (Infections and infestations) | 2 | 0 | NA | NA
Bacteraemia (Infections and infestations) | 1 | 1 | NA | NA
Biliary tract infection (Infections and infestations) | 1 | 0 | NA | NA
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | NA | NA
Candida infection (Infections and infestations) | 0 | 1 | NA | NA
Cellulitis (Infections and infestations) | 0 | 2 | NA | NA
Cerebral fungal infection (Infections and infestations) | 1 | 0 | NA | NA
Clostridial sepsis (Infections and infestations) | 1 | 0 | NA | NA
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | NA | NA
Clostridium difficile infection (Infections and infestations) | 0 | 1 | NA | NA
Coronavirus infection (Infections and infestations) | 1 | 0 | NA | NA
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | NA | NA
Device related infection (Infections and infestations) | 1 | 2 | NA | NA
Diverticulitis (Infections and infestations) | 0 | 1 | NA | NA
Enterococcal sepsis (Infections and infestations) | 1 | 1 | NA | NA
Gastroenteritis (Infections and infestations) | 0 | 1 | NA | NA
Gastroenteritis clostridial (Infections and infestations) | 1 | 0 | NA | NA
H1N1 influenza (Infections and infestations) | 1 | 0 | NA | NA
Hepatosplenic candidiasis (Infections and infestations) | 2 | 0 | NA | NA
Infection (Infections and infestations) | 0 | 2 | NA | NA
Kidney infection (Infections and infestations) | 1 | 0 | NA | NA
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | NA | NA
Klebsiella sepsis (Infections and infestations) | 1 | 0 | NA | NA
Neutropenic sepsis (Infections and infestations) | 3 | 1 | NA | NA
Pelvic abscess (Infections and infestations) | 1 | 0 | NA | NA
Pharyngeal abscess (Infections and infestations) | 0 | 1 | NA | NA
Pneumonia (Infections and infestations) | 9 | 12 | NA | NA
Pneumonia fungal (Infections and infestations) | 2 | 1 | NA | NA
Pneumonia viral (Infections and infestations) | 0 | 1 | NA | NA
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | NA | NA
Pulmonary sepsis (Infections and infestations) | 0 | 2 | NA | NA
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | NA | NA
Respiratory tract infection (Infections and infestations) | 1 | 0 | NA | NA
Sepsis (Infections and infestations) | 11 | 13 | NA | NA
Septic shock (Infections and infestations) | 8 | 9 | NA | NA
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | NA | NA
Streptococcal infection (Infections and infestations) | 1 | 0 | NA | NA
Streptococcal sepsis (Infections and infestations) | 3 | 0 | NA | NA
Systemic candida (Infections and infestations) | 0 | 2 | NA | NA
Systemic mycosis (Infections and infestations) | 0 | 1 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | NA | NA
Viral myocarditis (Infections and infestations) | 0 | 1 | NA | NA
Expired product administered (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Alanine aminotransferase increased (Investigations) | 1 | 1 | NA | NA
Aspartate aminotransferase increased (Investigations) | 0 | 1 | NA | NA
Body temperature increased (Investigations) | 0 | 1 | NA | NA
C-reactive protein increased (Investigations) | 1 | 0 | NA | NA
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 1 | NA | NA
Electrocardiogram QT prolonged (Investigations) | 0 | 2 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | NA | NA
Hepatic enzyme increased (Investigations) | 0 | 1 | NA | NA
Lymphocyte count increased (Investigations) | 0 | 1 | NA | NA
Neutrophil count decreased (Investigations) | 0 | 1 | NA | NA
Platelet count decreased (Investigations) | 0 | 3 | NA | NA
Pulmonary function test decreased (Investigations) | 1 | 0 | NA | NA
White blood cell count decreased (Investigations) | 0 | 1 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 2 | NA | NA
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Cytarabine syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | NA | NA
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | NA | NA
Cerebral infarction (Nervous system disorders) | 1 | 0 | NA | NA
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | NA | NA
Dizziness (Nervous system disorders) | 0 | 1 | NA | NA
Facial paresis (Nervous system disorders) | 0 | 1 | NA | NA
Facial spasm (Nervous system disorders) | 1 | 0 | NA | NA
Myelopathy (Nervous system disorders) | 0 | 1 | NA | NA
Somnolence (Nervous system disorders) | 1 | 0 | NA | NA
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | NA | NA
Syncope (Nervous system disorders) | 2 | 1 | NA | NA
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | NA | NA
Depression (Psychiatric disorders) | 0 | 1 | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 1 | NA | NA
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | NA | NA
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | NA | NA
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Embolism (Vascular disorders) | 1 | 0 | NA | NA
Hypotension (Vascular disorders) | 1 | 0 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Midostaurin + Chemotherapy (On-treatment) (N=245) | Placebo + Chemotherapy (On-treatment) (N=249) | Midostaurin + Chemotherapy (Post-treatment Survival Follow-up) (N=0) | Placebo + Chemotherapy (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 77 | 96 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 102 | 116 | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 20 | 31 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 34 | 53 | NA | NA
Pancytopenia (Blood and lymphatic system disorders) | 6 | 13 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 62 | 69 | NA | NA
Tachycardia (Cardiac disorders) | 14 | 16 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 41 | 46 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 24 | 34 | NA | NA
Constipation (Gastrointestinal disorders) | 77 | 84 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 121 | 142 | NA | NA
Dyspepsia (Gastrointestinal disorders) | 16 | 16 | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 27 | 18 | NA | NA
Nausea (Gastrointestinal disorders) | 141 | 137 | NA | NA
Neutropenic colitis (Gastrointestinal disorders) | 13 | 5 | NA | NA
Proctalgia (Gastrointestinal disorders) | 13 | 5 | NA | NA
Stomatitis (Gastrointestinal disorders) | 39 | 36 | NA | NA
Vomiting (Gastrointestinal disorders) | 101 | 63 | NA | NA
Asthenia (General disorders) | 17 | 15 | NA | NA
Chills (General disorders) | 16 | 11 | NA | NA
Fatigue (General disorders) | 36 | 26 | NA | NA
Mucosal inflammation (General disorders) | 47 | 50 | NA | NA
Oedema (General disorders) | 27 | 21 | NA | NA
Oedema peripheral (General disorders) | 44 | 38 | NA | NA
Pain (General disorders) | 15 | 8 | NA | NA
Pyrexia (General disorders) | 146 | 138 | NA | NA
Device related infection (Infections and infestations) | 9 | 16 | NA | NA
Folliculitis (Infections and infestations) | 16 | 4 | NA | NA
Pneumonia (Infections and infestations) | 32 | 29 | NA | NA
Sepsis (Infections and infestations) | 13 | 13 | NA | NA
Transfusion reaction (Injury, poisoning and procedural complications) | 13 | 11 | NA | NA
Alanine aminotransferase increased (Investigations) | 29 | 29 | NA | NA
Aspartate aminotransferase increased (Investigations) | 24 | 18 | NA | NA
Blood alkaline phosphatase increased (Investigations) | 9 | 13 | NA | NA
Blood bilirubin increased (Investigations) | 19 | 7 | NA | NA
C-reactive protein increased (Investigations) | 15 | 13 | NA | NA
Electrocardiogram QT prolonged (Investigations) | 26 | 13 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 17 | 26 | NA | NA
Neutrophil count decreased (Investigations) | 20 | 20 | NA | NA
Platelet count decreased (Investigations) | 34 | 50 | NA | NA
Weight increased (Investigations) | 17 | 24 | NA | NA
White blood cell count decreased (Investigations) | 25 | 35 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 31 | 40 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 14 | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18 | 16 | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 24 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 95 | 102 | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 16 | 20 | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 16 | 18 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 14 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 32 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 13 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 15 | NA | NA
Dizziness (Nervous system disorders) | 14 | 23 | NA | NA
Headache (Nervous system disorders) | 70 | 64 | NA | NA
Anxiety (Psychiatric disorders) | 9 | 15 | NA | NA
Insomnia (Psychiatric disorders) | 16 | 25 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 37 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 27 | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 44 | 43 | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 22 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 14 | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 8 | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 20 | 20 | NA | NA
Petechiae (Skin and subcutaneous tissue disorders) | 20 | 21 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 28 | 32 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 80 | 87 | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 17 | 21 | NA | NA
Hypertension (Vascular disorders) | 20 | 27 | NA | NA
Hypotension (Vascular disorders) | 17 | 25 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT03512197/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT03512197/SAP_001.pdf